CLINICAL TRIAL: NCT05981482
Title: Accuracy and Utility of the Oxford Visual Perception Screening (OxVPS), a Screening for Visual Perception Difficulties in Stroke Survivors
Brief Title: Visual Perception Difficulties After Stroke
Status: Recruiting | Type: Observational
Sponsor: Durham University (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); County Durham and Darlington NHS Foundation Trust (Other Government); University of Oxford (Other)
Responsible Party: Principal Investigator, Kate Cowen, Postdoc researcher, Durham University
Other Study IDs: Durham University
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Visual Perception
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stroke survivors: Individuals who have survived a stroke
  Interventions: Diagnostic Test: OxVPS

INTERVENTIONS:
Diagnostic Test: OxVPS — Comparing a new screening tool, the Oxford visual perception screening, to the gold standard, Rivermead Perceptual Battery Assessment.

SUMMARY:
The goal of this observational study is to learn how well the Oxford Visual Perception Screening (OxVPS) tool can identify stroke survivors with visual perception difficulties.

The main aim is to determine the accuracy and utility of the OxVPS compared to the current gold standard assessment in stroke survivors. In other words, how well can the Oxford Visual Perception Screening tool (OxVPS) identify stroke patients with visual perception problems?

Participants will completed the OxVPS and the current gold standards visual perception screening tool.

DETAILED DESCRIPTION:
This is a non-experimental cross-sectional study. It aims to compare the new screening test OxVPS to the gold standard tests for visual perception difficulties.

Patients will be recruited at stroke rehabilitation units at hospitals in the North East of England and in Oxfordshire.

Following consent:

* Participants will complete the paper version of the Oxford Visual Perception Screen OxVPS (~15 min).
* Participants will complete screening for visual perception problems with a validated screening tool (~30-120 min).
* Participants will complete screening for cognition alterations and sensory vision with validated screening tools. (~30 min)
* Stroke details (time since stroke, severity) and demographic data (age, socio-economic status) will be collected to evaluated representativeness of the sample.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of stroke (ischemic stroke and/or intracerebral haemorrhage).
* Within 6 weeks of confirmed stroke.

Exclusion Criteria:

* Insufficient understanding of English
* Clinical concerns that patient is unable follow simple instructions.
* Clinical concerns that patient is unable to concentrate for 15 minutes.
* No capacity to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors on stroke rehabilitation units in the North East of England and Oxfordshire.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Validity of OxVPS | All testing completed in 2 weeks
  Convergent and discriminate validity will be assessed. Convergent validity expressed as a correlation between total score on OxVPS and RPAB. Discriminate validity to be expressed as correlation between OxVPS score and scores of cognitive and sensory vision assessments. Both calculated by a non-parametric Spearman correlation and estimate a 95% confidence interval. The analysis can be completed through the cor.test function in the base package of R.
Reliability of OxVPS | 2 weeks
  The inter-rater reliability of OxVPS will be evaluated through a Bland-Altman analysis [26]: we will calculate the difference in OxVPS scores between raters for each patient. Subsequently, we will plot the difference in scores as a function on the average score to evaluate a bias between the raters (mean difference) that might vary based on severity of a patient's visual perceptual problems. We will report the mean difference, standard deviation, and limits of agreement within where 95% of differences between raters fall. A t-test will indicate if the mean difference is significantly different from 0. Analyses will be performed in R with the functions from blandr package (e.g. blandr.statistics and blandr.draw) or functions from a similar package.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Vancleef, PhD, Principal Investigator — Durham University
Locations (3):
- United Kingdom (3):
  - Abingdon Community Hospital, Abingdon
  - Bishop Auckland Hospital, Bishop Auckland
  - Queen Elizabeth Hospital, Gateshead

IPD SHARING:
Plan to Share IPD: No